CLINICAL TRIAL: NCT03611686
Title: Observatory of Patients With Metastatic ProstAte Adenocarcinoma That is Resistant to Castration and Multi-LinE Strategies
Acronym: OPALE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/090/HP
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Prostate Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient followed for metastatic prostate adenocarcinoma: patient wil be followed for metastatic prostate adenocarcinoma during 3 years
  Interventions: Drug: Local chemotherapy

INTERVENTIONS:
Drug: Local chemotherapy — Local chemotherapy will be administrated according to local recommendation

SUMMARY:
Evaluation the overall survival of patients with metastatic prostate adenocarcinoma resistant to castration

ELIGIBILITY:
Inclusion Criteria:

* Patient monitored for castration-resistant metastatic prostate
* Patients starting a first or second line treatment as part of castration resistance
* Patient not objecting to the study after reading the information letter
* Patient aged over 18 years

Exclusion Criteria:

* Patient monitored for non-metastatic prostate cancer
* Patient monitored for castration-nonresistant prostate cancer
* Patient not able to understand the information letter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic prostate adenocarcinoma resistant to castration
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of alive patient | 3 years

SECONDARY OUTCOMES:
Number of alive patient disease free | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian PFISTER, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No